CLINICAL TRIAL: NCT02654626
Title: A Randomized, Single-blind, Placebo-controlled, Sequential Parallel-Group and Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability and Pharmacokinetics of KBP-7072 in Healthy Subjects
Brief Title: A Multiple Ascending Dose Study of KBP-7072 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KBP Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KBP7072-1-002
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — kbp-7072

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- KBP-7072: Cohort 1 (Experimental): Healthy Volunteers will receive multiple dose of KBP-7072 and placebo
  Interventions: Drug: KBP-7072; Other: Placebo
- KBP-7072: Cohort 2 (Experimental): Healthy Volunteers will receive multiple dose of KBP-7072 and placebo
  Interventions: Drug: KBP-7072; Other: Placebo
- KBP-7072: Cohort 3 (Experimental): Healthy Volunteers will receive multiple dose of KBP-7072 and placebo
  Interventions: Drug: KBP-7072; Other: Placebo
- KBP-7072: Cohort 4 (Experimental): Healthy Volunteers will receive multiple dose of KBP-7072 and placebo
  Interventions: Drug: KBP-7072; Other: Placebo

INTERVENTIONS:
Drug: KBP-7072 — Drug Intervention
Other: Placebo

SUMMARY:
This is a randomized, single-blind, placebo-controlled, sequential parallel-group and multiple ascending dose (MAD) study to evaluate the safety, tolerability and pharmacokinetics of KBP 7072 in healthy subjects. The safety will be assessed at each dose level before progressing to the next higher dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject
* Are between the ages of 18 and 55 years (inclusive);
* Body mass index (BMI) of 19 to 30 kg/m2 inclusive and body weight not less than 50 kg.

Exclusion Criteria:

* Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity;
* Known or suspected malignancy;
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody;
* Positive pregnancy test result.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (i.e., number of participants with adverse events, abnormal vital signs, clinical laboratory findings, 12-lead ECGs and physical examinations) in healthy subjects | up to 17 days

SECONDARY OUTCOMES:
Area Under Curve (AUC) in healthy subjects | up to 10 days
  on Day 1 (first dose): pre-dose (within 30 minutes prior to dosing) and 0.5, 1, 2, 4, 6, 10, 12, 18, and 24 hours post dose; on Days 4, 7, 8, and 9: pre-dose (within 30 minutes prior to dosing); on Day 10 (last dose): pre-dose (within 30 minutes prior to dosing) and 0.5, 1, 2, 4, 6, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Laboratories, Inc., Secaucus, New Jersey, United States

REFERENCES:
- [Derived] Huband MD, Mendes RE, Pfaller MA, Lindley JM, Strand GJ, Benn VJ, Zhang J, Li L, Zhang M, Tan X, Liu Q, Flamm RK. In Vitro Activity of KBP-7072, a Novel Third-Generation Tetracycline, against 531 Recent Geographically Diverse and Molecularly Characterized Acinetobacter baumannii Species Complex Isolates. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02375-19. doi: 10.1128/AAC.02375-19. Print 2020 Apr 21. PMID 32071042